CLINICAL TRIAL: NCT07176507
Title: MULTIVALVE : A Prospective Multicentre Study of Multiple and Mixed Valvular Heart Disease
Acronym: MULTIVALVE
Status: Not yet recruiting | Type: Observational
Sponsor: French Cardiology Society (Other)
Responsible Party: Sponsor
Other Study IDs: 2023-A02626-39
Record Dates: First submitted 2025-07-24; First posted 2025-09-16 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Valvular Heart Disease
Keywords: valvular heart disease; Multiple and mixed valvular heart disease; multiple valve disease
MeSH Terms: conditions — Heart Valve Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples Without DNA — optional blood sample <56ml
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with a diagnosis of MMVD: Patients with a diagnosis of MMVD based on cardiovascular imaging and defined as follows:
  At least two cases of moderate to severe valvular heart disease, as assessed by a cardiologist and defined by transthoracic echocardiography (TTE) on one or more valves. This is in line with the recommendations of the European Society of Cardiology (ESC), the American Society of Echocardiography (ASE) and expert opinion.

SUMMARY:
Multiple and mixed valvular heart disease (MMVD) is a common condition in clinical practice. It corresponds to a combination of stenotic or leaky lesions on two or more heart valves (multiple valve disease), or a combination of stenotic and leaky lesions on the same valve (mixed valve disease). However, the management of their clinical, biological and cardiovascular imaging is not well established. Current European Society of Cardiology (ESC) recommendations primarily address the various valve diseases in isolation. This results in an absence of reliable recommendations for managing MMVD, with different approaches being adopted by care centres.

In order to address this knowledge gap regarding MMVD, it is crucial to assess its prevalence, the cardiovascular imaging methods employed and the management strategies, as well as to identify prognostic factors for the various combinations of valve disease.

The multicentre MMVD study will be a valuable resource as it will improve our understanding of the prognosis for patients with MMVD. It will highlight imaging and biological markers associated with the prognosis of different combinations of MMVD.

DETAILED DESCRIPTION:
National, Prospective, Multicentric Registry. Patients with a diagnosis of MMVD identified by echocardiography will be included and followed up at 1, 2, 3 and 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* The patient has been informed of the study and has not refused to participate.
* An echocardiographic diagnosis of MMVD is defined as having at least two moderate to severe valvulopathies, as assessed by a cardiologist using transthoracic echocardiography (TTE), on one or more valves. This is in line with the recommendations of the ESC, the ASE, and expert opinion.

Exclusion Criteria:

* History of valve surgery or percutaneous valve intervention involving the valve in question.
* A history of infective endocarditis, whether treated surgically or not, confirmed according to the modified Duke criteria.
* Acute infective endocarditis at the time of evaluation for inclusion, confirmed according to the modified Duke criteria.
* Complex congenital heart disease.
* Patients who are already included in the European EACVI-MMVD study.
* Pregnant women
* Patients not affiliated to social security
* Patients who are minors
* Patients under guardianship, curatorship or judicial supervision
* Patients who refuse to participate in this register.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a diagnosis of MMVD based on cardiovascular imaging and defined as follows:
  At least two cases of moderate to severe valvular heart disease, as assessed by a cardiologist and defined by transthoracic echocardiography (TTE) on one or more valves. This is in line with the recommendations of the European Society of Cardiology (ESC), the American Society of Echocardiography (ASE) and expert opinion.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2025-10 (Estimated); Primary Completion 2028-10 (Estimated); Study Completion 2032-10 (Estimated)

PRIMARY OUTCOMES:
To assess the association between cardiovascular imaging parameters (echocardiography and/or cardiac MRI) and cardiovascular event-free survival in a population of MMVD. | 1 year after inclusion
  Survival without cardiovascular event

SECONDARY OUTCOMES:
To assess the association between cardiovascular imaging parameters and survival | at 1, 2, 3 and 5 years after inclusion
Proportion of patients who did not experience a cardiovascular event | at 1, 2, 3 and 5 years after inclusion
Proportion of patients who are alive | at 1, 2, 3 and 5 years after inclusion
Proportion of patients who did not experience a cardiovascular event depending on the type of treatment (medical, surgical or percutaneous) | at 1, 2, 3 and 5 years after inclusion
Proportion of patients who are alive depending on the type of treatment (medical, surgical or percutaneous) | at 1, 2, 3 and 5 years after inclusion
To assess the progression of the stage of severity of valvulopathy | at 1, 2, 3 and 5 years after inclusion
  Echocardiography
% of patients with MMVD combinations | during 5 years after inclusion
Measurement of cardiovascular biomarkers | at baseline and 1, 2, 3 and 5 years after inclusion
  BNP or NT-pro-BNP and troponin
Assessing the association between cardiovascular biomarkers in patients with MMVD and survival | during 5 years after inclusion
  BNP or NT-pro-BNP and troponin, vital status
Assessing the association between cardiovascular biomarkers in patients with MMVD and cardiovascular event-free survival | during 5 years after inclusion
  BNP or NT-pro-BNP and troponin, Survival without cardiovascular event
Exploring the value of cardiovascular biomarkers analysed in a centralised laboratory (optional) | at baseline
  Biobank (optional)

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Chu Lille- Hopital Cardiologique, Lille
  - Chu Lariboisiere (Aphp), Paris

IPD SHARING:
Plan to Share IPD: Undecided